CLINICAL TRIAL: NCT00485745
Title: Repeat Sternotomy for Pediatric Cardiac Surgery: Indications, Risks and Results
Brief Title: Repeat Sternotomy for Pediatrics
Status: Completed | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Sponsor
Other Study IDs: 07-023
Record Dates: First submitted 2007-06-12; First posted 2007-06-13 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Congenital Disorders
Keywords: surgery; repeat sternotomy; pediatrics
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Given the relative lack of information regarding the risks associated with repeat sternotomy in the pediatric patient population, a preliminary screen of the Children's Cardiothoracic Surgery Database was performed to determine how many repeat sternotomies have been performed at this institution within the last 4 years. A total of 1281 repeat sternotomies were identified during this time period.

We propose a retrospective review of the indications, potential risk factors, and short-term outcomes for these procedures. These data would allow a multivariable regression analysis to identify risk factors associated with adverse events during repeat sternotomy.

DETAILED DESCRIPTION:
Median sternotomy is the most common approach for cardiac surgery in adults and children. While the initial sternotomy is rarely associated with adverse events, the risks associated with repeated sternotomies for subsequent reoperations may be higher. This increased risk is primarily due to adhesions securing cardiac structures to the sternum, thus placing those structures at risk for injury during sternal re-entry. There have been several large studies examining the frequency and impact of adverse events during repeat sternotomy in adults. Roselli and colleagues from the Cleveland Clinic reviewed 1853 consecutive repeat sternotomies and found a 6.8% incidence of serious adverse events. 1 This study can be contrasted against the report of O'Brien and colleagues which reviewed the results of 546 repeat sternotomies performed over 21 years in Brisbane, Australia with only 9 (1.6%) minor cardiac injuries and no major adverse events. 2

The pediatric cardiac surgical field is somewhat different from the adult realm in that re-operations are more common, either due to planned, staged palliation requiring multiple operations or the expected failure of implanted conduits and valves which subsequently require replacement. However, while the incidence of repeat sternotomy is higher in the pediatric population, the overall number of patients is considerably smaller, so there has been a relative dearth of information in the literature regarding the risks and outcomes associated with repeat sternotomy. The largest series reported was published by Russell and colleagues in 1998 and included only 192 repeat sternotomies performed on 165 patients. 3 The authors reported a 5.2% incidence of cardiac laceration with selective utilization of femoro-femoral bypass to decompress the heart during repeat sternotomy for "higher risk" patients.

ELIGIBILITY:
Inclusion Criteria:

* Repeat sternotomy at Children's Healthcare of Atlanta between 1.1.02 and 12.31.06
* patient under 21 years of age
* "repeat" is defined as a sternotomy performed more than 1 month after the most recent previous sternotomy

Exclusion Criteria:

* Those charts that do not meet inclusion criteria

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population for this retrospective chart review will be all patients, under 21 years of age who have undergone a repeat sternotomy at Children's Healthcare of Atlanta at Egleston between January 1, 2002 and December 31, 2006. A repeat sternotomy is defined as having been performed more than a month after the most recent previous sternotomy.
Sampling Method: Probability Sample
Enrollment: 1281 (Actual)
Dates: Start 2002-01; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Retrospective medical record review evaluating preoperative and intraoperative variables associated with repeat sternotomy as risk factors for adverse events. | Length of stay
  This study will be a retrospective medical record review evaluating preoperative and intraoperative variables associated with repeat sternotomy as risk factors for adverse events. Short-term outcomes including ventilator time, intensive care unit and hospital length of stay, blood product utilization, and transfusions will be analyzed to determine the effect of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Kirshbom, MD, Principal Investigator — Children's Healthcare of Atlanta